CLINICAL TRIAL: NCT06592586
Title: A Follow-up Trial to Assess the Persistence of the Immune Response to the Group B Streptococcus Vaccine (GBS-NN/NN2) After a Primary Vaccination of Healthy Pregnant Women, and to Assess Safety, Reactogenicity, and Immunogenicity of the GBS-NN/NN2 Vaccine When Administered During Follow-Up as a 1 Booster Dose During a New Pregnancy
Brief Title: A Follow-up Trial of GBS-NN/NN2 Vaccine in Healthy Pregnant Women
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Minervax ApS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MVX008; 2024-516364-28 (EudraCT Number)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Streptococcus Agalactiae Infection; Neonatal Sepsis; Pneumonia; Meningitis; Neonatal Infection; Gram-Positive Bacterial Infections; Bacterial Infections; Bacterial Infections and Mycoses; Infections
Keywords: Immunology; Streptococcus agalactiae; Lancefield's Group B Streptococcus; Pregnancy
MeSH Terms: conditions — Streptococcal Infections; Neonatal Sepsis; Pneumonia; Meningitis; Gram-Positive Bacterial Infections; Bacterial Infections; Bacterial Infections and Mycoses; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Non-Pregnant Participants: No GBS-NN/NN2 Booster Dose (No Intervention): Participants who received at least one dose of GBS-NN/NN2 during the parent studies but do not become pregnant during this study will not receive the GBS-NN/NN2 booster dose.
- Pregnant Participants: GBS-NN/NN2 Booster Dose (Experimental): Participants who received at least one dose of GBS-NN/NN2 during the parent studies and, become pregnant during this study, and qualify, will receive become pregnant during this study will receive the GBS-NN/NN2 booster dose.
  Interventions: Biological: GBS-NN/NN2 vaccine
- Pregnant Participants: No GBS-NN/NN2 Booster Dose (No Intervention): Participants who received at least one dose of GBS-NN/NN2 during the parent studies and, become pregnant during this study but do not qualify for receiving the GBS-NN/NN2 booster dose.

INTERVENTIONS:
Biological: GBS-NN/NN2 vaccine — 0.5 mL (50 μg GBS-NN +50 μg GBS-NN2 adsorbed to 0.5 mg aluminium as Alhydrogel®)
  Arms: Pregnant Participants: GBS-NN/NN2 Booster Dose

SUMMARY:
The main objective of the study is to evaluate the persistence of the immunoglobulin G (IgG) antibody responses, specific to Alpha-like protein CN (AlpCN), Ribosomal Protein N (RibN), Alpha-like protein 1N (Alp1N), and Alpha-like protein 2 and 3 (Alp2-3N), after a primary vaccination with GBS-NN/NN2 in all participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant living in Denmark or South Africa who has participated either in Trial MVX0004 (NCT05154578) or MVX0005 (NCT04596878) and has received at least 1 dose of the GBS-NN/NN2 vaccine.
* Participant who is able to read and understand and capable of giving personal signed informed consent.
* Participant who is willing and able to comply with scheduled visits, the investigational plan, and other trial procedures.
* Participant who is granting access to their trial-related medical records and to their trial materials from Trials MVX0004 or MVX0005, whatever is applicable.
* Participant who are expected to be available for the duration of the trial and who can be contacted by telephone during trial participation.

Exclusion Criteria:

* Any personnel involved in the conduct of the trial (and their family members), including, but not limited to, site staff members, MinervaX employees, and any vendor or contract research organisation (CRO) employees.
* Participant with confirmed Group B Streptococcus (GBS) infection since participation in Trial MVX0004 or MVX0005.
* Participant with any psychiatric condition, including recent (within the past year) active suicidal ideation/behaviour that may increase the risk of trial participation or, in the investigator's judgement, make the participant unsuitable for participation in the trial.
* Participant who participated in other trials involving investigational drug(s) or devices within 28 days prior to trial entry, and/or are participating in other trials involving investigational drug(s) or devices at trial entry, or plan to (continue to) participate in other trials involving investigational drug(s) or devices during this trial.
* Participant with known or suspected immunodeficiency or cancer or a family history of congenital or hereditary immunodeficiency.
* Participant receiving chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to trial entry. An immunosuppressive dose of glucocorticoid will be defined as a systemic dose ≥10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
* Participant who received blood, blood products, plasma derivatives, or any immunoglobulin preparations in the 12 weeks prior to trial entry or is planning to receive such products during this trial.
* Participant with current or history of drug or alcohol abuse, as judged by the investigator.
* Participant who received any marketed or investigational (other than GBS-NN/NN2 in the MVX0004 or MVX0005 Trial) GBS vaccines or who is planning to receive any marketed or investigational (other than GBS NN/NN2) GBS vaccines during this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
All Participants: Concentration of IgG Antibodies to AlpN Proteins in Blood Serum | Up to approximately 5 years

SECONDARY OUTCOMES:
Concentration of IgG Antibodies to AlpN Proteins in Blood Serum Following GBS-NN/NN2 Booster Dose | Pre-dose, 1 month pots-dose, at delivery, and 6 months post-delivery
Difference in Concentration of IgG Antibodies Between Maternal and Cord Blood at Delivery Following GBS-NN/NN2 Booster Dose | Up until delivery, approximately 5 years
Concentration of IgG Antibodies to AlpN Proteins in Blood Serum at Delivery in the Absence of GBS-NN/NN2 Booster Dose | Up until delivery, approximately 5 years
Difference in Concentration of IgG Antibodies Between Maternal and Cord Blood at Delivery in the Absence of GBS-NN/NN2 Booster Dose | Up until delivery, approximately 5 years
Concentration of IgG Antibody to AlpN Proteins in Blood Serum of Offspring from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | At delivery and at 1 and 3 months post-birth
Concentration of IgG Antibody to AlpN Proteins in Cord Blood of Offspring from Pregnant Participants who did not Received the GBS-NN/NN2 Booster Dose | Up until birth, approximately 5 years
All Participants: Number of Participants Experiencing Procedure-related Serious Adverse Events (SAEs) | Up to approximately 5 years
Number of Participants Experiencing Solicited Local and Systemic Adverse Events (AEs) Among Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up to approximately Day 7
Number of Participants Experiencing Unsolicited AEs Among Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up to approximately Day 28
Number of Participants Experiencing SAEs Among Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up to approximately 6 months post-delivery
Number of Participants Experiencing AE of Special Interest (AESI) Among Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up until delivery, approximately 5 years
Gestational Age (GA) of Offspring from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up until birth, approximately 5 years
Weight of Offspring from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up until birth, approximately 5 years
Length of Offspring from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up until birth, approximately 5 years
Head Circumference of Offspring from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up until birth, approximately 5 years
Apgar Score of Offspring from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up until birth, approximately 5 years
Number of Offspring Experiencing Unsolicited AEs from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up to 1 month post-birth, approximately 5 years
Developmental Milestones of Offspring from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose as Assessed by the Ages & Stages Questionnaire, 3rd Edition (ASQ-3) | At 6 months post-birth, approximately 5 years
Number of Offspring Experiencing Medically-attended AEs (MAAEs) from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up to 6 months post-birth, approximately 5 years
Number of Offspring Experiencing SAEs from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up to 6 months post-birth, approximately 5 years
Number of Offspring Experiencing AESIs from Pregnant Participants who Received the GBS-NN/NN2 Booster Dose | Up to 6 months post-birth, approximately 5 years

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (3):
  - Hvidovre Hospital - Department Of Obstetrics And Gynaecology, Copenhagen, Capital Region
  - Aarhus Universitetshospital, Aarhus N, Central Jutland
  - Sygehus Lillebælt - Kolding Sygehus, Kolding, Region Syddanmark
- South Africa (3):
  - Sefako Makgatho Health Sciences University, Medunsa Clinical Research Unit (MeCRU), Ga-Rankuwa, Gauteng
  - Wits Reproductive Health and HIV Institute (Wits RHI), Johannesburg, Guateng Province
  - Setshaba Research Centre, Pretoria, Guateng Province